CLINICAL TRIAL: NCT00003455
Title: Phase II Study of Oral Antineoplastons A10 and AS2-1 in Women With Advanced Breast Cancer
Brief Title: Antineoplaston Therapy in Treating Women With Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BC-BR-14; CDR0000066487 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Stage IV Breast Cancer; Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1; Biological Therapy; Complementary Therapies

INTERVENTIONS:
Drug: antineoplaston A10
Drug: antineoplaston AS2-1
Procedure: alternative product therapy
Procedure: biological therapy
Procedure: biologically based therapies
Procedure: cancer prevention intervention
Procedure: complementary and alternative therapy
Procedure: differentiation therapy

SUMMARY:
RATIONALE: Antineoplastons are naturally-occurring substances that may also be made in the laboratory. Antineoplastons may inhibit the growth of cancer cells.

PURPOSE: This phase II trial is studying how well antineoplaston therapy works in treating women with stage IV breast cancer that has not responded to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of antineoplastons A10 and AS2-1 capsules in patients with advanced breast cancer by determining the proportion of women who experience an objective tumor response.
* Evaluate the adverse effects of and tolerance to this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive oral antineoplaston A10 and antineoplaston AS2-1 6 to 7 times per day.

Treatment continues for at least 6 weeks. Patients achieving complete or partial response may continue on therapy until disease progression or toxic effects occur.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV breast cancer that is unlikely to respond to existing therapy and for which no curative therapy exists
* Failed prior standard therapy
* Measurable disease by MRI or CT scan
* Tumor must be at least 2 cm in the lymph nodes in the head, neck, axillary, inguinal, or femoral areas and at least 0.5 cm in other locations
* Hormone receptor status:
* Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal Status:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal failure

Cardiovascular:

* No chronic heart failure
* No uncontrolled hypertension

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious medical or psychiatric disorders
* No active infections
* No other serious concurrent disease
* No serious malabsorption syndromes

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from prior immunotherapy
* At least 4 weeks since prior immunotherapy, except in patients with disease progression during or after initial therapy

Chemotherapy:

* Recovered from prior chemotherapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas), except in patients with disease progression during or after initial therapy

Endocrine therapy:

* Recovered from prior hormonal therapy
* At least 12 weeks since prior hormonal therapy, except in patients with disease progression during and after initial therapy
* Concurrent corticosteroids for peritumoral edema allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered
* Patients with multiple tumors who have received radiotherapy to some, but not all, tumors may be admitted earlier than 8 weeks

Surgery:

* Recovered from any prior surgery
* No prior extensive stomach or intestinal surgery

Other:

* Prior cytodifferentiating agents allowed
* No prior antineoplaston therapy
* No other concurrent therapy for metastatic breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States